CLINICAL TRIAL: NCT02238158
Title: Postmarketing Surveillance (as Per §67(6)AMG [German Drug Law]) of Atrovent® in Chronic Obstructive Pulmonary Disease
Brief Title: Postmarketing Surveillance of Atrovent® in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 244.2496
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease
  Interventions: Drug: Atrovent® inhalets

INTERVENTIONS:
Drug: Atrovent® inhalets

SUMMARY:
To obtain further information on the tolerability and efficacy of Atrovent® inhalets in long term treatment of Chronic Obstructive Pulmonary Disease under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Primarily patients of both gender, older than 40 years, who suffer from Chronic Obstructive Pulmonary Disease
* Only patients who had not been treated with Atrovent® within the last year were to be considered for inclusion

Exclusion Criteria:

• Contraindications listed in the Instructions for Use/Summary of Product Characteristics for Atrovent® Inhalets

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive airways disease recruited at general practitioners
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 1999-09; Primary Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Investigator assessment of improvement of the clinical picture rated on a 6-point symptom profile | Up to 12 months after first study drug administration

SECONDARY OUTCOMES:
Assessment of efficacy by investigator on a 4-point scale | Up to 12 months after first study drug administration
Assessment of efficacy by patient on a 4-point scale | Up to 12 months after first study drug administration
Assessment of tolerability by investigator on a 4-point scale | Up to 12 months after first study drug administration
Assessment of tolerability by patient on a 4-point scale | Up to 12 months after first study drug administration
Number of patients with adverse drug reactions | Up to 12 months after first study drug administration